CLINICAL TRIAL: NCT07025928
Title: Salt Intake and Blood Pressure Control in Adults With Essential Hypertension
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Jingfeng (Other)
Responsible Party: Sponsor-Investigator, Sun Jingfeng, Family Physician, SingHealth Polyclinics
Organization: SingHealth Polyclinics (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-0006; SHP-CG-CRGNov24-A05 (Other: SingHealth Polyclinic Collaborative Research Grant)
Record Dates: First submitted 2025-04-03; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Hypertension; sodium reduction; increased potassium intake; reduced salt; blood pressure control; primary care; Singapore; educational intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be masked to group allocation. While both groups will receive educational materials, participants in the control arm will not be informed that the Patient Information Leaflet (PIL) is the comparator intervention. This design minimizes expectancy bias by ensuring participants are unaware of whether they are receiving the "active" DSHP Diet Tool or the control material. Outcome assessors analyzing biochemical and clinical data will also be masked to group allocation to reduce detection bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DSHP Diet Tool and DSHP Patient information leaflet (Experimental): Participants in this arm will receive standard hypertension care along with access to the Decreased Salt High Potassium (DSHP) Diet Tool for 24 weeks and DSHP Patient information leaflet. The DSHP Tool is a patient-centered educational resource developed to support sodium reduction and increase potassium intake through practical strategies, goal setting, and food guidance. Participants will also receive the DSHP Patient Information Leaflet (PIL). Patients will be guided on how to use the tool by a study coordinator. Clinical and dietary assessments will be conducted at baseline and at the end of the intervention.
  Interventions: Behavioral: Decreased Salt High Potassium Tool (DSHP Tool)
- Standard Care + DSHP Patient Information Leaflet (No Intervention): Participants in this arm will receive standard hypertension care as provided at SingHealth Polyclinics, along with the DSHP Patient Information Leaflet (PIL). The PIL provides written guidance on reducing sodium and increasing potassium intake. No access to the DSHP Tool will be provided in this arm. Participants will undergo the same clinical and dietary assessments as the intervention group at baseline and after 24 weeks.

INTERVENTIONS:
Behavioral: Decreased Salt High Potassium Tool (DSHP Tool) — Participants in this arm will receive standard hypertension care and the Decreased Salt High Potassium (DSHP)Tool for 24 weeks. The DSHP Tool is an educational resource which includes a sodium intake calculator and tracker, potassium-rich food lists, risk matrix visuals, goal-setting modules tailored to the Singaporean diet. Participants will also receive the DSHP Patient Information Leaflet (PIL) .
  Arms: DSHP Diet Tool and DSHP Patient information leaflet

SUMMARY:
The goal of this study is to explore the barriers and facilitators to adopting a reduced dietary salt and increased potassium intake among adults with essential hypertension in Singapore, and to evaluate the feasibility and preliminary effectiveness of a newly developed educational tool-Decreased Salt High Potassium (DSHP) Diet Tool-in reducing dietary sodium intake and increasing potassium intake.

This three-part study will involve adults aged 21 years and above, with a self-reported diagnosis of hypertension for at least six months and/or currently taking antihypertensive medication. Participants will be recruited from two SingHealth Polyclinics (Punggol Polyclinic and Pasir Ris Polyclinic). Healthcare providers (HCPs) working at these clinics who have experience in managing patients with hypertension and in educating patients on reducing dietary sodium intake will also be recruited.

The main questions this study aims to answer are:

* What are the perceived barriers and facilitators for patients with hypertension to reduce dietary sodium and increase potassium intake?
* What are the perceived barriers and facilitators experienced by healthcare providers in educating patients about sodium reduction and potassium intake?
* Is the DSHP Diet Tool feasible and effective in reducing dietary sodium intake and increasing potassium intake among patients with hypertension?

Participants in the intervention group will be provided DSHP Diet Tool and Decreased Salt High Potassium patient information leaflet (DSHP PIL). Participants in the control group will receive standard care and a patient information leaflet (DSHP PIL). Researchers will compare participants in the intervention group to the control group to determine whether the DSHP tool is effective in reducing dietary sodium and increasing potassium intake in patients with hypertension.

DETAILED DESCRIPTION:
Hypertension is a major public health concern globally, contributing to cardiovascular disease and premature mortality. According to the World Health Organization (2023), one in three adults worldwide suffers from hypertension. In Singapore, the 2022 National Population Health Survey reported that over 35% of residents aged 18 to 74 years had hypertension, with nearly 65% of those under medical follow-up exhibiting poor blood pressure control. One of the most significant and modifiable risk factors for hypertension is diet-specifically, excessive sodium (salt) intake and insufficient potassium intake.

Excess sodium elevates blood pressure by causing fluid retention and adversely affecting vascular function. Conversely, potassium intake helps regulate blood pressure through mechanisms like promoting sodium excretion and reducing vascular resistance. The benefits of dietary sodium reduction and increasing potassium intake are well-established in both clinical trials and population studies, particularly in individuals with hypertension.

Despite this, Singaporeans continue to consume well above the recommended daily intake for sodium and below the optimal levels for potassium. The average sodium intake is approximately 3,620 mg/day (exceeding the WHO recommendation of 2,000 mg/day), while potassium intake averages 2,500 mg/day (below the recommended 3,510 mg/day). Public health initiatives like the "War on Salt" campaign (launched in 2011) have had limited long-term success in addressing these dietary gaps.

Previous studies in Singapore and neighboring countries have identified significant gaps in knowledge, attitudes, and behaviors related to dietary sodium and potassium. However, there has been limited research focused on practical, context-specific educational interventions aimed at improving dietary behaviors related to salt and potassium intake, especially within the hypertensive population in the primary care setting.

Study Objectives and Hypothesis This study is designed in three parts to systematically develop, refine, and evaluate a novel educational tool-the Decreased Salt High Potassium (DSHP) Diet Tool-for hypertensive patients. The tool aims to support patients in reducing dietary sodium and increasing potassium intake, thereby improving blood pressure control and overall cardiovascular risk profiles.

Primary Hypothesis: A targeted educational tool, developed based on patient and healthcare provider input, will be feasible and effective in supporting reductions in sodium intake and increases in potassium intake among hypertensive patients, leading to improved blood pressure outcomes.

Objectives:

Part 1:

* Identify perceived barriers, facilitators, and attitudes towards reduced sodium and increased potassium diets among hypertensive patients.
* Understand healthcare providers' (HCPs) perspectives on the barriers in educating patients about reducing sodium intake and increasing potassium intake.

Part 2:

* Develop a prototype DSHP Diet Tool based on findings from Part 1.
* Alpha-test the tool with both patients and HCPs to assess usability and acceptability.
* Refine the tool through multiple feedback cycles using qualitative interviews and usability surveys (System Usability Scale - SUS).

Part 3:

* Conduct a pilot randomized controlled trial (RCT) to evaluate the feasibility, usability, and preliminary effectiveness of the DSHP Diet Tool in real-world clinical settings.

Study Design Overview

The study will be conducted in three distinct but interrelated parts:

Part 1: Qualitative study

Design: Qualitative study using in-depth interviews and/or focus group discussions guided by the Theoretical Domains Framework (TDF). Population: 40 hypertensive patients and 20 healthcare providers from two SingHealth Polyclinics (Punggol and Pasir Ris). Sampling: Purposive sampling to ensure diversity in age, gender, ethnicity in patients Data Collection:

* Audio-recorded, semi-structured interviews will be carried out Data Analysis: Thematic analysis using the TDF as a guiding framework. Coding will be conducted independently by multiple researchers to ensure reliability. Data collection will continue until saturation is achieved.

Part 2: Development and Alpha Testing of DSHP Diet Tool

Design: Mixed-methods developmental study. Tool Development: Content developed using findings from Part 1 and validated through collaboration with dietitians, nurses, content experts, and HCPs. Components include:

* General education on sodium and potassium.
* Sodium intake calculator and tracker.
* Food lists and risk matrix.
* Behavior change strategies and goal setting.
* Progress tracking and support resources.

Alpha Testing:

* 20 hypertensive patients and 20 HCPs will test the tool over four iterative cycles (5 patients and 5 HCPs per round).
* Participants will use the DSHP Tool for two weeks.
* Feedback collected via System Usability Scale (SUS) and semi-structured interviews.
* DSHP Tool will be revised based on feedback from each cycle.

Outcome Measures:

* SUS scores (target usability score ≥ 68).
* Feedback on usability and feasibility of the DSHP Tool

Part 3: Pilot Randomized Controlled Trial (RCT) Design: Parallel, two-arm, 1:1 allocation pilot RCT with mixed-method evaluation. Sites: SingHealth Polyclinic - Punggol and SingHealth Polyclinic - Pasir Ris. Sample Size: 80 patients with hypertension (40 per arm), with 25% over-recruitment to account for attrition. Randomization: Using sealed, sequentially numbered opaque envelopes (SNOEs) prepared by an independent researcher. Duration: 24-week intervention period.

Arms:

* Intervention Group: DSHP Tool + Patient Information Leaflet (PIL).
* Control Group: Standard care + PIL.

Assessments (Baseline and 24 weeks):

* Blood pressure (systolic/diastolic)
* Body weight and height
* Serum sodium, potassium, creatinine
* 24-hour urinary sodium and potassium
* Salt literacy and DASH adherence scores

Qualitative Component: At the end of the RCT, a subset of patients from the intervention group will participate in interviews to provide in-depth feedback on acceptability, usability of the DSHP Tool.

Statistical Methods

Quantitative Analysis:

* Independent t-tests or Wilcoxon rank-sum tests for group comparisons.
* Paired t-tests or Wilcoxon signed-rank tests for within-group comparisons.
* Categorical variables analyzed using chi-square tests.
* Intention-to-treat (ITT) principles will be used.
* Missing data managed via multiple imputation or last observation carried forward.

Qualitative Analysis:

* Framework analysis based on TDF.
* Coding verified by multiple investigators.
* Triangulation with quantitative data for integrated interpretation.

Ethical Considerations and Safety

* The study has obtained approval from the SingHealth Centralised Institutional Review Board (CIRB).
* Written informed consent will be obtained from all participants.
* Participants may withdraw at any time without penalty.
* All data will be de-identified and stored securely.
* Risks include potential discomfort during interviews or dietary changes, and rare risks such as hyperkalemia or hyponatremia. Patients at risk of hyperkalemia or hyponatremia are excluded from participation.

Expected Impact and Significance

This study aims to address critical gaps in dietary management of hypertension in Singapore by:

* Developing a practical, theory-informed, user-centered dietary tool.
* Empowering patients to self-manage their hypertension through improved dietary habits.
* Supporting HCPs with an effective educational resource.

ELIGIBILITY:
Inclusion Criteria for patients:

* Participants who are 21 years old and above.
* Participants who self-reports to have hypertension for at least six months and/ or taking at least one type of antihypertensive medication daily for at least six months
* Able to read English

Exclusion Criteria for patients:

* Participants with type 1/ type 2 or secondary diabetes mellitus
* Participants with CKD stage 3B and above
* Participants with serum potassium of above 4.5mmol/L (on the latest blood test)
* Participants with serum sodium of less than 135 mmol/L (on the latest blood test)
* Participants who are on daily potassium chloride
* Participants who are on diuretics (thiazide or thiazide like diuretics)
* Participants who are pregnant
* Participants who had been diagnosed with any terminal illnesses, visually impaired, disability or mental health related illnesses (visually impaired refers to individuals who self-report to have difficulty reading the wordings on the patient consent form, even with the use of visual aids)
* Participants who are not clinically stable (Clinically stable patients are defined in this study as:
* Has clinic BP 100-160/60-100 mmHg, Heart Rate (HR) 60-100 bpm
* No recent hospitalizations (within the last 3 months) due to hypertensive emergencies, strokes, myocardial infarctions or other acute cardiovascular events
* No recent symptoms such as severe dizziness, fainting, or chest pain) *Participants who are on PRN potassium supplements is not an exclusion criteria

Inclusion criteria for Healthcare providers:

* HCPs who had prior experience in advising patients on dietary salt reduction
* HCPs who self-reported to have ever treated patients with hypertension

Exclusion criteria for healthcare providers

-nil

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
24 hour Urinary Sodium level | At baseline and at the end of the intervention (24 weeks)
  24 hour urinary sodium level will be assessed at baseline and at the end of the intervention
24 hour urinary potassium level | at baseline and at the end of intervention (24 weeks)
  24 hour urinary potassium level will be measured at baseline and at the end of intervention (24 weeks)

SECONDARY OUTCOMES:
Blood pressure | at baseline and at the end of intervention (24 weeks)
  Blood pressure will be assessed at baseline and at the end of the intervention (24 weeks)
Body mass index | at baseline and at the end of 24 weeks
  Body mass index will be measured at baseline and at the end of 24 weeks
Salt literacy scale | At baseline and at the end of intervention (24 weeks)
  Salt literacy scale will be measured at baseline and at the end of intervention (24 weeks). Changes in salt literacy will be assessed using a validated Health Literacy Scale for Low Salt Consumption, which measures participants' knowledge, attitudes, and behaviors related to salt intake. The salt literacy scale has a possible score ranging from 0 to 98, with a higher score indicating higher health literacy related to low salt intake.
DASH score | at baseline and at the end of intervention (24 weeks)
  DASH score will be measured at baseline and at the end of intervention (24 weeks). Adherence to the DASH (Dietary Approaches to Stop Hypertension) diet will be evaluated using the DASH score questionnaire, reflecting overall dietary behavior in relation to sodium and potassium intake. Minimum Score: 0, Maximum Score: 63 , with higher score indicating better adherence to the DASH diet

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns about maintaining participant confidentiality and data privacy. As the study involves sensitive health information and is conducted in a clinical setting, data sharing could increase the risk of re-identification despite de-identification measures. Additionally, participants were not consented for public data sharing at the time of enrollment.

REFERENCES:
- [Background] Silva-Santos T, Moreira P, Rodrigues M, Padrao P, Pinho O, Norton P, Ndrio A, Goncalves C. Interventions That Successfully Reduced Adults Salt Intake-A Systematic Review. Nutrients. 2021 Dec 21;14(1):6. doi: 10.3390/nu14010006. PMID 35010883
- [Background] Cheong SM, Ambak R, Othman F, He FJ, Salleh R, Mohd Sallehudin S, Palaniveloo L, Ganapathy SS. Knowledge, perception, and practice related to sodium intake among Malaysian adults: findings from the Malaysian Community Salt Study (MyCoSS). J Health Popul Nutr. 2021 May 31;40(Suppl 1):5. doi: 10.1186/s41043-021-00231-4. PMID 34059162
- [Background] Chan CMJ, Dickens BSL, Chong MF. Understanding knowledge, attitudes and behaviours related to dietary sodium intake in a multi-ethnic population in Singapore. Public Health Nutr. 2023 Dec;26(12):2802-2814. doi: 10.1017/S1368980023002422. Epub 2023 Nov 3. PMID 37921207
- [Background] Aaron KJ, Sanders PW. Role of dietary salt and potassium intake in cardiovascular health and disease: a review of the evidence. Mayo Clin Proc. 2013 Sep;88(9):987-95. doi: 10.1016/j.mayocp.2013.06.005. PMID 24001491
- [Background] Ekmekcioglu C, Elmadfa I, Meyer AL, Moeslinger T. The role of dietary potassium in hypertension and diabetes. J Physiol Biochem. 2016 Mar;72(1):93-106. doi: 10.1007/s13105-015-0449-1. Epub 2015 Dec 3. PMID 26634368
- [Background] Koh J, Ang G, Tan KB, Chen C. The social cost of high sodium diet in Singapore. Br J Nutr. 2023 May 14;129(9):1598-1606. doi: 10.1017/S0007114522001568. Epub 2022 May 26. PMID 35614498
- [Background] Bibbins-Domingo K, Chertow GM, Coxson PG, Moran A, Lightwood JM, Pletcher MJ, Goldman L. Projected effect of dietary salt reductions on future cardiovascular disease. N Engl J Med. 2010 Feb 18;362(7):590-9. doi: 10.1056/NEJMoa0907355. Epub 2010 Jan 20. PMID 20089957
- [Background] Pimenta E, Gaddam KK, Oparil S, Aban I, Husain S, Dell'Italia LJ, Calhoun DA. Effects of dietary sodium reduction on blood pressure in subjects with resistant hypertension: results from a randomized trial. Hypertension. 2009 Sep;54(3):475-81. doi: 10.1161/HYPERTENSIONAHA.109.131235. Epub 2009 Jul 20. PMID 19620517
- [Background] He FJ, Li J, Macgregor GA. Effect of longer-term modest salt reduction on blood pressure. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD004937. doi: 10.1002/14651858.CD004937.pub2. PMID 23633321
- [Background] Grillo A, Salvi L, Coruzzi P, Salvi P, Parati G. Sodium Intake and Hypertension. Nutrients. 2019 Aug 21;11(9):1970. doi: 10.3390/nu11091970. PMID 31438636
- [Background] Adrogue HJ, Madias NE. Sodium and potassium in the pathogenesis of hypertension. N Engl J Med. 2007 May 10;356(19):1966-78. doi: 10.1056/NEJMra064486. No abstract available. PMID 17494929
- [Background] Vaduganathan M, Mensah GA, Turco JV, Fuster V, Roth GA. The Global Burden of Cardiovascular Diseases and Risk: A Compass for Future Health. J Am Coll Cardiol. 2022 Dec 20;80(25):2361-2371. doi: 10.1016/j.jacc.2022.11.005. Epub 2022 Nov 9. No abstract available. PMID 36368511